CLINICAL TRIAL: NCT05162391
Title: Effects of Methamphetamine Use on Risk Behavior, Systemic and Mucosal Inflammation, and Sexually Transmitted Infection (STI)/HIV Risk Among Men Who Have Sex With Men
Brief Title: Inflammation in Methamphetamine and STIs (IMSTI)
Acronym: IMSTI
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Cherie Blair, MD, PhD, Assistant Clinical Professor, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DA054004-01A1
Record Dates: First submitted 2021-11-30; First posted 2021-12-17 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Methamphetamine-dependence; Rectal Gonorrhea; Rectal Chlamydia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Contingency management (Other): All enrolled participants will participate in a Contingency Management intervention where rewards are linked with demonstrated abstinence from methamphetamine use.
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management intervention with incentives tied to provision of urine samples with no detectable levels of methamphetamine (MA).

SUMMARY:
This clinical trial aims to investigate the effects of a decline in methamphetamine use on rectal inflammatory cytokine levels, substance use contexts, and HIV/STI risk behavior. This clinical trial also seeks to evaluate joint effects of methamphetamine use and rectal gonorrhea/chlamydia infection on rectal inflammatory cytokine levels. The proposed trial will consist of 40 MSM, half with rectal gonorrhea/chlamydia infection at enrollment (n=20), with methamphetamine use disorder that will receive contingency management for methamphetamine reduction. Following baseline measurement, participants will be observed over the course of 8 weeks, where participants will complete behavioral surveys, provide urine for drug testing, and rectal samples for measurement of rectal inflammatory cytokine levels.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender male
* 18 years of age or older
* Understand written and spoken English
* Condomless receptive anal intercourse in past 90 days
* Meet DSM-5 criteria for methamphetamine use disorder
* Positive urine toxicology screen for MA metabolites at study entry
* Negative rectal GC/CT screen (n=20) or Positive rectal GC and/or CT screen (n=20)
* Able to provide written informed consent and willing/able to complete study visits.

Exclusion Criteria:

* Reports current treatment for another substance use disorder
* Positive test for opioids, cocaine, and/or hallucinogens
* Treatment for gonorrhea and/or chlamydia infection in past 3 months
* Presence of a condition that in the opinion of the investigator would compromise the safety of the patient or the quality of the data

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Methamphetamine abstinence | 8 weeks
  Proportion of visits in which there are no detectable methamphetamine metabolites in participant urine samples
Rectal inflammation | 8 weeks
  Rectal concentrations of IL-6 (pg/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Cherie Blair, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Vine Street Clinic, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided